CLINICAL TRIAL: NCT06003621
Title: A Single Arm, Open-label, Phase II Signal-seeking Trial of Tiragolumab and Atezolizumab in Patients With Advanced Solid Tumours.
Brief Title: Tiragolumab and Atezolizumab in Advanced Pan-cancer Patients
Acronym: MoST-TAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Omico (Other)
Collaborators: Hoffmann-La Roche (Industry); The George Institute for Global Health, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML43743
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Tiragolumab; atezolizumab

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, single-arm, open-label, phase II signal-seeking trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tiragolumab and atezolizumab (Experimental): 96 patients will be treated with tiragolumab for one cycle (600mg IV over 60-90 minutes). At Cycle 2 Day 1, participants receive IV tiragolumab (600mg) and atezolizumab (1,200mg) over 60-90 minutes. Cycles of tiragolumab and atezolizumab repeat every 21 days, with infusion time decreased (if tolerable) until treatment discontinuation, with or without disease progression.
  Because of the heterogeneity of eligible cancer types, and lack of knowledge about relevant cut-offs for this combination, analysis will be performed prospectively to allocate patients into 4 subgroups based on the following tumour characteristics;
  * Group 1: TMB ≥ 10, assessed using NGS panel screening. n=24
  * Group 2:Tumour and immune cell PD-L1 expression (TAP score) > 20% high or PD-L1 (CD274) amplification, defined as gene copy number > 6 on the panel. n=24
  * Group 3: Tumour and immune cell PD-L1 expression (TAP score) 5% - 20% int. n=24
  * Group 4: Tumour infiltrating lymphocytes CD3+CD8+ ≥ 5%. n=24
  Interventions: Biological: Tiragolumab; Biological: Atezolizumab

INTERVENTIONS:
Biological: Tiragolumab — 600mg IV every 21 days from Cycle 1 Day 1
  Other Names: RO7092284; MTIG7192A; RG-6058; Anti-TIGIT
Biological: Atezolizumab — 1,200mg IV every 21 days from Cycle 2 Day 1
  Other Names: Tecentriq; MPDL3280A; RG7446; RO5541267

SUMMARY:
This phase II study will explore the effect of 2 monoclonal antibodies, tiragolumab and atezolizumab, in patients with locally advanced solid cancers which cannot be removed by surgery or have spread. Their cancers will have characteristics which may predict immune response to the study treatment. PD-L1 and TIGIT are immune receptors which can help cancers grow by evading the immune response and inhibiting the action of some immune cells. By blocking these receptors, tiragolumab and atezolizumab may work together to re-activate the body's anti-tumour immune response and kill cancer cells.

DETAILED DESCRIPTION:
Patients who are enrolled in the MoST or CaSP cancer screening programs, and whose tumour is assessed as amenable to tiragolumab and atezolizumab treatment, will be recommended for participation in the study. After being informed about the study, and the potential risks, patients who consent to participate undergo a 21-day screening period to determine study eligibility. Patients will be prospectively selected into subgroups based on their tumour characteristics.

Once eligibility is confirmed, tiragolumab alone is administered at Cycle 1 Day 1 (day 1 of study). Commencing from Cycle 2 Day 1, tiragolumab and atezolizumab are administered at 21-day cycles until treatment discontinuation, with or without disease progression.

Participants undergo a biopsy at cycle 2 prior to commencement of atezolizumab treatment. Standard imaging scans (usually computed tomography (CT)) are performed throughout the trial. Patients also undergo blood, urine and stool sample collection on study.

Once participants discontinue treatment, a study visit is performed within 30 days of the end of the final treatment cycle. If treatment cessation is not contemporaneous with disease progression, follow-up calls are conducted every 9 weeks until disease progression. Once disease progression occurs, a study visit is performed within 30 days of disease progression and then every 3 months until 12 months after the final participant discontinues study treatment.

Active follow-up of all participants will continue until death or 12 months after the last participant discontinues study treatment, whichever occurs first. Subsequently, survival data will be obtained through MoST or CaSP until death.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Aged ≥18 years old.
3. Histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumour.
4. Exhausted all available standard therapy or not suitable for standard therapy (including targeted therapies) for the tumour.
5. ECOG performance status score of 0-1.
6. Sufficient and accessible tumour tissue for panel sequencing, PD-L1 and TIL testing, and tertiary objectives.
7. Tumour biomarker criteria predictive of immune response defined by presence of one or more of the following;

   * Group 1: tumour mutation burden ≥ 10 mutations per megabase.
   * Group 2: PD-L1 amplification >6 copy number alterations
   * Group 3: tumour PD-L1 expression TAP score ≥ 5%
   * Group 4: tumour infiltrating lymphocytes (TILs) (CD3+CD8+) ≥ 5%.
8. Patient is willing to provide tumour biopsy samples on treatment at Week 4.
9. Life expectancy >12 weeks.
10. Measurable disease as defined by iRECIST or RANO criteria.
11. Adequate haematological and biochemical indices as defined by:

    * Absolute neutrophil count ≥1.0 x 10^9/L
    * Haemoglobin ≥100 g/L
    * Platelet count ≥100 x 10^9/L
    * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5x ULN; or ≤5.0x ULN if liver metastases are present.
    * International normalised ratio (INR) <1.3 in the absence of anticoagulation therapy.
    * Serum creatinine clearance >40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance.
12. Negative HIV test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy, have a CD4 count ≥ 200cells/mm3 , and have an undetectable viral load.
13. Negative hepatitis B surface antigen (HBsAg) test at screening.
14. Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

    * Negative total hepatitis B core antibody (HBcAb);
    * Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL.

    The HBV DNA test must be performed for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
15. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test must be performed for patients who have a positive HCV antibody test.
16. Women of childbearing potential must have a negative screening serum pregnancy test within 14 days prior to the first dose of study medication.
17. Women of childbearing potential and men must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the study and for at least 5 months after the last dose of study medication.
18. Ability to adhere to the study visit schedule and understand and comply with all protocol requirements and instructions from study staff.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Roche staff and/or staff at the study site).
2. Patients with non-small cell lung cancer.
3. Participation in another clinical study with an investigational product during the last 4 weeks prior to study enrolment.
4. Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
5. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
6. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-α [TNF-α] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

   * topical, intranasal, or inhaled corticosteroids or systemic corticosteroids at or below physiological doses (eg. ≤10 mg/day of prednisone);
   * use of dexamethasone up to 4mg/day within 14 days of initial treatment for patients with brain tumours.
7. Symptomatic or actively progressing central nervous system (CNS) metastases.

   Asymptomatic patients with treated or untreated CNS lesions are eligible, provided that all of the following criteria are met:
   * Measurable disease, per RECIST v1.1, must be present outside the CNS.
   * The patient has no history of intracranial haemorrhage or spinal cord haemorrhage.
   * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
   * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease.
   * If the patient is receiving anti-convulsant therapy, the dose is considered stable.
   * Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
   * There is no evidence of interim progression between completion of CNS directed therapy (if administered) and initiation of study treatment.

   Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy and/or surgery, with no need to repeat the screening brain scan.
8. Prior use of approved or investigational anti-TIGIT therapy.
9. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
10. Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives prior to initiation of study treatment.
11. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
12. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      i. Rash must cover < 10% of body surface area; ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids; and iii. There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
13. Active or prior documented inflammatory bowel disease requiring systemic treatment within the past 2 years (e.g., Crohn's disease, ulcerative colitis).
14. History of primary immunodeficiency.
15. History of allogeneic organ transplant.
16. History of hypersensitivity to mAb to PD1/PD-L1 or any excipient.
17. Uncontrolled intercurrent illness including, but not limited to:

    * Ongoing or active infection
    * Symptomatic congestive heart failure
    * Uncontrolled hypertension
    * Unstable angina pectoris
    * Cardiac arrhythmia
    * Active peptic ulcer disease or gastritis
    * Active bleeding diatheses
    * Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrolment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

    Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy, if appropriate, prior to enrolment.
    * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX®) are allowed.
    * Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected calcium greater than ULN)
    * Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
18. Active tuberculosis.
19. Positive EBV viral capsid antigen (VCA) IgM test during screening. An EBV polymerase chain reaction (PCR) test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
20. History of leptomeningeal carcinomatosis.
21. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
22. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
23. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving tiragolumab and atezolizumab.
24. Pregnant or breastfeeding.
25. Contraindication to study treatments as judged by the patient's responsible clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate at 6 Months | 6 months
  The primary outcome, PFS rate at 6 months, is defined as the proportion of participants who are alive and progression free at 6 months from start of study treatment
  Radiological disease progression is defined according to modified Response Evaluation Criteria in Solid Tumours version 1.1 for immune-based therapeutics (iRECIST) or Response Assessment in Neuro-Oncology criteria (RANO).
  Clinical progression is defined as the development of:
  1. Symptoms attributable to cancer progression; or
  2. Initiation of other anticancer treatment for cancer; or
  3. Significant deterioration of performance status not explained by treatment toxicities, co-morbidities, or radiological evidence of progression; or
  4. Unequivocal development of new non-measurable disease that is not assessable according to iRECIST or RANO criteria.

SECONDARY OUTCOMES:
Objective tumour response rate (OTRR) as per iRECIST or RANO criteria | iRECIST/RANO every 9 weeks from study entry to objective disease progression, up to 18 months
  The objective tumour response rate is defined as the proportion of participants who achieved an objective response at any time point.
  Participants with an objective tumour response are defined as those assessed as having a complete or partial response according to iRECIST or RANO. Investigator assessed response status (i.e. complete response, partial response, stable disease or progressive disease) will be assessed by using iRECIST or RANO at each assessment time point. Confirmation of progressive disease will be undertaken in accordance to the iRECIST criteria.
The median duration of objective tumour response | iRECIST/RANO every 9 weeks from study entry to objective disease progression, up to 18 months
  Median duration of objective tumour response is defined as the time interval from documentation of an objective tumour response to date of first evidence of radiological disease progression.
Median PFS | iRECIST/RANO every 9 weeks from study entry to objective disease progression, up to 60 months
  PFS is defined as the interval from the start date of study treatment to the date of first evidence of disease progression (clinical or radiological) or death from any cause, whichever occurs first.
  Median PFS will be calculated. Participants who did not progress or who are still alive will be censored on the date of their last clinical assessment or tumour assessment.
To evaluate the duration of clinical benefit (DCB) | iRECIST/RANO every 9 weeks from study entry to objective disease progression, up to 60 months
  DCB is defined as the time interval from date of start of study treatment to date of first evidence of radiological disease progression.
To evaluate the overall survival (OS) rate at 12 months | Cycle 1 Day 1 to 12 months
  OS is defined as the interval from the start date of study treatment to date of death from any cause. Participants who did not die will be censored at the date of last known follow-up alive.
  OS rate at 12 months is defined as the proportion of participants who are alive at 12 months, from start date of study treatment to date of death from any cause (or the date of last known vital status during follow up within 12 months from start date of study treatment).
To calculate the median overall survival | Cycle 1 Day 1 to death, up to 5 years
  Median OS will be calculated
To evaluate the time to progression (TTP) | iRECIST/RANO every 9 weeks from study entry to objective disease progression, up to 60 months
  TTP is defined as the time interval from the start date of study treatment to the date of first evidence of disease progression on the MoST-TAP trial or death due to cancer.
To calculate the median Growth Modulation Index (GMI) | iRECIST/RANO every 9 weeks from study entry to objective disease progression, up to 60 months
  To assess clinical benefit while taking into account the disease tempo of individual patients, GMI, defined as the ratio of TTP using tiragolumab and atezolizumab in the MoST-TAP trial with the TTP in the period prior to MoST-TAP, will be calculated. GMI estimates the duration of clinical benefit normalised against the disease tempo, as estimated by the TTP before enrolment onto the MoST-TAP trial.
  If GMI is ≥1.3, then the study therapy will be defined as having benefit for the participant. The median GMI will be calculated.
The incidence and rates of AEs and serious AEs (SAEs) | From Cycle 1 Day 1 to 90 days after cessation of study drug
  The safety and tolerability of tiragolumab and atezolizumab treatment will be assessed by the incidence and rates of AEs and serious AEs (SAEs). AEs will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
  Tolerability is defined as the time from commencement of study treatment until interruption of treatment due to toxicity. Interruption of treatment includes treatment discontinuation or a pause in treatment. Toxicity is defined as a treatment-related AE equal to or above Grade 3 as graded by CTCAE v5.0. An AE is deemed to be due to treatment if the causal relationship between the event and tiragolumab or atezolizumab treatment is judged by the Investigator to be definitely, probably or possibly related.
To evaluate the health related quality of life (HRQOL) over the course of the trial | Cycle 1 Day 1, Cycle 4 Day 1 and then every third cycle until disease progression (cycles length 21 days). Also administered at the Treatment Discontinuation Visit and the Progressive Disease Visit.
  HRQOL will be measured by the EORTC Quality of Life of Cancer Patients (QLQ-C30 v3).
  The questionnaire includes functional, symptom and global health status / QoL scales. Patients rate items on the questionnaire from 1 (not at all) to 4 (very much) or from 1 (very poor) to 7 (excellent).
  Questionnaires are administered at Cycle 1 Day 1 (baseline, Week 1), Cycle 4 Day 1 (Week 10) and then every 3 cycles until disease progression. Questionnaires are also administered at the Treatment Discontinuation Visit and the Progressive Disease Visit.

CONTACTS AND LOCATIONS:
Overall Officials: David Thomas, PHD, FRACP, Principal Investigator — Omico; UNSW Sydney
Locations (13):
- Australia (13):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Ramsay Health Care Australia Pty Ltd trading as The Border Cancer Hospital, Albury, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Orange Base Hospital, Orange, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Health, Bendigo, Victoria
  - Barwon Health, Geelong, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided
Subject to further IRB review and protocol amendment